CLINICAL TRIAL: NCT05567731
Title: Effect of Long, Short, and Ultrashort GnRH Agonist Treatment Protocols in Intracytoplasmic Sperm Injection Candidates on Ovarian Reserve
Brief Title: Effect of GnRH Agonist Treatment Protocols on Ovarian Reserve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Ossman, Assistant Professor of Obstetrics and Gynecology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35416/4/22
Record Dates: First submitted 2022-10-02; First posted 2022-10-05 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Intracytoplasmic Sperm Injection; GnRH Agonist; Infertility; Ovarian Reserve
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ultrashort GnRHa (Experimental): the patients used the ultrashort protocols with GnRH agonist (GnRH-a, and recombinant FSH for controlled ovarian hyperstimulation (COH). Form the second day of menstrual cycle, 0.1 mg/d GnRH agonist will be injected by subcutaneous injection for 3-4 d.
  Interventions: Drug: ultrashort GnRHa
- short GnRHa (Experimental): Buserelin acetate 100 mg five times daily and FSH will be started on the 2nd day of the menstrual cycle as short application. The dose of gonadotropin hormone will be individualized according to the patient's age and previous stimulation history or response to stimulation. Cycles will be monitored by transvaginal ultrasonography and serum E2 levels.
  Interventions: Drug: short GnRHa
- long GnRHa (Experimental): In the long protocol, daily SC injection of Triptorelin :Decapeptyl 0.1 mg (Ferring, Switzerland) 0.1 mg started at day 21 of the cycle prior to stimulation cycle and continued till the day of hCG triggering. Gn stimulation started after fulfilling stimulation start criteria of thin endometrium < 5 mm and low E2 < 50 and LH < 5IU/l with either HMG(Menogon; Ferring, Switzerland) or rFSH (Gonal-f; Merck Serono, Germany) in a starting dose of 150-300 IU/day according to women age, day 3 FSH,AMH and previous gonadotropin response then adjustment of the dose according to ovarian response monitored by serum E2 and ultrasound evaluation. All patients were followed up by Transvaginal ultrasound scan daily or on alternate days according to the ovarian response to treatment starting on treatment cycle day for folliculometry and endometrial thickness and pattern.
  Interventions: Drug: long GnRHa

INTERVENTIONS:
Drug: ultrashort GnRHa — the patients used the ultrashort protocols with GnRH agonist (GnRH-a, and recombinant Follicle-Stimulating Hormone for controlled ovarian hyperstimulation (COH). Form the second day of menstrual cycle, 0.1 mg/d GnRHa will be injected by subcutaneous injection for 3-4 d.
  Gonadotropins will be added from the third day of menstrual cycle and the initial gonadotropin doses will be 225-300 IU/d. During the treatment, gonadotropin doses will be adjusted according to guided monitoring of follicle growth and measurement of serum estradiol (E2) levels of 10 000 units of human chorionic gonadotrophin (hCG) will be administered when 43 follicles will be 418 mm
  Other Names: ultrashort gonadotropin-releasing hormone (GnRH) agonist
  Arms: ultrashort GnRHa
Drug: short GnRHa — Buserelin acetate 100 mg five times daily and FSH will be started on the 2nd day of the menstrual cycle as short application. The dose of gonadotropin hormone will be individualized according to the patient's age and previous stimulation history or response to stimulation. Cycles will be monitored by transvaginal ultrasonography and serum estradiol (E2) levels.
  Follicular maturation will be completed by the administration of 10000 IU human chorionic gonadotrophin (hCG) when at least two follicles reached a diameter of >18 mm. Thirty-five to thirty-six hours after human chorionic gonadotrophin (hCG) administration, ovum retrieval will be performed by transvaginal echo-guided ovarian puncture.
  Other Names: short gonadotropin-releasing hormone (GnRH) agonist
  Arms: short GnRHa
Drug: long GnRHa — In the long protocol, daily subcutaneuous injection of Triptorelin :Decapeptyl 0.1 mg (Ferring, Switzerland) 0.1 mg started at day 21 of the cycle prior to stimulation cycle and continued till the day of hCG triggering. Gn stimulation started after fulfilling stimulation start criteria of thin endometrium < 5 mm and low estradiol (E2) < 50 and Luteinizing Hormone < 5IU/l with either HMG(Menogon; Ferring, Switzerland) or rFSH (Gonal-f; Merck Serono, Germany) in a starting dose of 150-300 IU/day according to women age, day 3 Follicle-Stimulating Hormone, Anti-Müllerian Hormone and previous gonadotropin response then adjustment of the dose according to ovarian response monitored by serum estradiol (E2) and ultrasound evaluation.
  Other Names: long gonadotropin-releasing hormone (GnRH) agonist
  Arms: long GnRHa

SUMMARY:
This study aimed to compare the gonadotropin-releasing hormone agonist (ultra-short) protocol versus (short and long) protocols on ovarian reserve in women undergoing intracytoplasmic sperm injection

DETAILED DESCRIPTION:
Infertility affects about 15% of all the couples attempting to generate pregnancy, of which can be attributed to female and male factors. For females, advanced age and poor ovarian reserve were the main causes which resulted in infertility.

Pituitary down-regulation with gonadotropin-releasing hormone (GnRH) agonists followed by ovarian stimulation with exogenous gonadotropins has been successfully used as standard hormonal treatment in women undergoing assisted reproductive technologies (ART) for the last 10 years. Ovulation induction is a frequently utilized therapeutic procedure for the management of infertility.

With the use of gonadotropin-releasing hormone agonists in controlled ovarian hyperstimulation (COH) protocols, the results of the ART improved in terms of reduction in cycle cancellation by the almost abolition of spontaneous LH surges (<2%). The GnRHa also reduce inadequate follicular development and imprecise clinical pregnancy rate.

Intracytoplasmic sperm injection (ICSI), it has allowed successful pregnancies and proved to be a consistent treatment for the alleviation of infertility due to severe semen abnormalities including cryptozoospermia.

ELIGIBILITY:
Inclusion Criteria:

* women
* aged between 18- and 35-years old
* undergoing Intracytoplasmic sperm injection.

Exclusion Criteria:

* History of three or more previous In vitro fertilisation failures
* Karyotypic abnormalities in either partner
* Patients who previously undergo unilateral oophorectomy
* Patients with chronic diseases (uncontrolled diabetes mellitus, cardiovascular diseases, liver and kidney failure)
* Patients with diseases may affect In vitro fertilisation outcomes (Endometriosis, uterine fibroids, Hydrosalpinx, Adenomyosis, autoimmune diseases), polycystic ovary syndrome (PCOS) patients, poor responders (maternal age >40, Antral follicle counts (AFC)<5, Anti Mullerian Hormone (AMH)<1 and previous trial <5 oocyte retrieved)
* Severe male factor, uterine abnormalities, adenomyosis and endometriosis
* History of malignant tumors and related treatment, clinically significant systemic disease or abnormal hematology, chemistry, or urinalysis results at screening, non-ovarian causes (male or tubal factors with average ovarian reserve).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women aged between 18- and 35-years old women undergoing Intracytoplasmic sperm injection
Enrollment: 30 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancies | 12 weeks postintervention
  Number of ongoing pregnancies per woman randomized, defined as evidence of a gestational sac with fetal heart motion at 12 weeks or later, confirmed with ultrasound.

SECONDARY OUTCOMES:
retrieved oocytes | 4 days postintervention
  Number of oocytes retrieved per woman randomized
Estradiol level | second day of menstruation
  Estradiol level will be recorded
Luteinizing Hormone level | second day of menstruation
  Luteinizing Hormone level will be recorded
Follicle-Stimulating Hormone level | second day of menstruation
  Follicle-Stimulating Hormone level will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed M.E. Ossman, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available under a reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: One year after the end of the study